CLINICAL TRIAL: NCT03594448
Title: Detection of Microsatellite Instability (MSI) in Circulating Tumor DNA of Patients With Stage IV Colorectal Carcinoma
Brief Title: Detection of MSI in Circulating Tumor DNA of Colorectal Carcinoma Patients
Status: Terminated | Type: Observational
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 3C-18-2; NCI-2018-01169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-18-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Microsatellite Instability; Colorectal Cancer Stage IV
MeSH Terms: conditions — Microsatellite Instability; Colorectal Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-correlative (Specimen collection): Participants undergo collection of blood samples in addition to the usual amount collected when they come in for their regular cancer treatments or doctor?s appointment every 6-8 weeks until disease progression or stopping at 9 months.
  Interventions: Procedure: Specimen Collection; Procedure: Serial Liquid Biopsy

INTERVENTIONS:
Procedure: Specimen Collection — Undergo collection of blood samples
Procedure: Serial Liquid Biopsy — Undergo serial liquid biopsy

SUMMARY:
This pilot trial studies how well serial liquid biopsies work in detecting microsatellite instability in participants with stage IV colorectal cancer. Serial liquid biopsies may help doctors learn better methods to track cancer in the bloodstream and how to use these to improve cancer treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that there is high level of concordance between the electrophoretic mobility profile of microsatellite biomarkers in circulating cell-free deoxyribonucleic acid (ccfDNA) versus in primary tumor tissues in patients with colorectal carcinomas displaying microsatellite instability.

II. To test the hypothesis that changes in the electrophoretic mobility profile of microsatellite biomarkers in liquid biopsies from patients with colorectal carcinoma correlate with therapeutic responsiveness measured based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

III. To determine whether microsatellite alleles generated as a result of microsatellite instability detectable in liquid biopsy specimens from patients with colorectal carcinoma represent the entire cancer cell population or only a subset of cancer cells differentially affected by genomic instability.

OUTLINE:

Participants undergo collection of blood samples to evaluate microsatellite instability via serial liquid biopsies at baseline, then every 6 weeks and at progression or 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with stage IV colorectal cancer and with defined microsatellite instability status before initiation of systemic immunotherapy.
* Trackable cancer-driver mutation in the primary tumor documented before initiation of chemotherapy.
* Zubrod performance status of 0 or 1.
* Patients have measurable disease according to RECIST version (v)1.1.
* Ability to understand and willing to sign a written informed consent.

Exclusion Criteria:

* Severe anemia (hemoglobin [Hb] < 8 g/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with stage IV colorectal cancer and with defined microsatellite instability status before initiation of systemic immunotherapy will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Correlation between presence of MSI present in circulating tumor DNA versus in primary tumor specimens | Up to 1 year
  MSI testing distinguishes between tumors into one of 3 phenotypic categories: MSI-High (MSI-H) is reported when > 30% of biomarkers show instability; Microsatellite stable (MSS) is reported in the absence of instability. The third category, MSI-Low (MSI-L) is diagnostically equivalent to MSS, and is reported when MSI is present in < 30% of biomarkers. MSI status will be determined by polymerase chain reaction (PCR) using commercial kits provided by Promega.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Josef Lenz, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California